CLINICAL TRIAL: NCT00424580
Title: Airway Responses to Montelukast and Desloratadine.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Saskatchewan (Other)
Responsible Party: Dr. Donald W. Cockcroft, Department of Medicine, University of Saskatchewan
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: BIO-REB# 06-232
Record Dates: First submitted 2007-01-18; First posted 2007-01-19 (Estimated); Last update posted 2008-01-23 (Estimated); Status verified 2008-01

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — montelukast; desloratadine

INTERVENTIONS:
Drug: Montelukast (10mg) and Desloratadine (5mg)

SUMMARY:
Montelukast (for asthma) and desloratadine (for allergies) are effective therapy for their current uses. Part of what happens when your allergies trigger your asthma should be prevented by either of these drugs. This project is being conducted to determine if these drugs are effective, either alone or in combination, on controlling asthma that is triggered by allergies.

ELIGIBILITY:
Inclusion Criteria:

* baseline FEV1 > or = 65% predicted
* positive methacholine challenge (i.e. methacholine PC20 < or = 16mg/ml
* positive allergen challenge

Exclusion Criteria:

* negative skin prick test
* lung condition/disease other than asthma
* currently use montelukast and/or desloratadine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12
Dates: Start 2007-01; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Late asthmatic response (maximum percent decrease in FEV1)

SECONDARY OUTCOMES:
Early asthmatic response (maximum percent decrease in FEV1
Changes in sputum cell/mediator content
Changes in airway hyperresponsiveness (methacholine PC20)

CONTACTS AND LOCATIONS:
Overall Officials: Donald W Cockcroft, MD, FRCP(C), Principal Investigator — University of Saskatchew Full Professor
Locations (1):
- Room 346 Ellis Hall, Saskatoon, Saskatchewan, Canada

REFERENCES:
- [Derived] Davis BE, Illamperuma C, Gauvreau GM, Watson RM, O'Byrne PM, Deschesnes F, Boulet LP, Cockcroft DW. Single-dose desloratadine and montelukast and allergen-induced late airway responses. Eur Respir J. 2009 Jun;33(6):1302-8. doi: 10.1183/09031936.00169008. Epub 2009 Jan 22. PMID 19164343